CLINICAL TRIAL: NCT05315388
Title: Effects of "Vitamin N" Nature Immersion Therapy on Stress Levels in Health Care Workers in the City of Bogotá: an Intervention Evaluation Study, 2022 - 2024.
Brief Title: Effects of "Vitamin N" Nature Immersion Therapy on Stress Levels in Health Care Workers in the City of Bogotá
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeadran N. Malagón-Rojas (Other Government)
Responsible Party: Sponsor-Investigator, Jeadran N. Malagón-Rojas, Coordinator, Grupo de Salud Ambiental Laboral, Principal Investigator, Medicine, Msc, PhD(c), Instituto Nacional de Salud, Colombia
Organization: Instituto Nacional de Salud, Colombia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-2021
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cortisol Excess; Stress, Psychological; Anxiety; Epigenetic Disorder; Natural Killer Cell Cytokine Production; Environmental Exposure
Keywords: Forest therapy; Nature therapy; Cortisol; Psychological stress; Physiological stress; Anxiety; Blood pressure; Natural Killer; DNA Methylation
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Stress, Psychological; Anxiety Disorders | interventions — Forest Therapy

STUDY DESIGN:
Intervention Model Description: Parallel intervention evaluation study that will consider two interventions; the conscious immersion therapy in nature (Vitamin N) and the usual intervention designed by the company for psychosocial risk reduction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1. Regular therapy group (No Intervention): Group without intervention during the study period no changes will be made in their daily routine. They will receive a weekly intervention operationalized for psychosocial risk.
- Group 2A: Vitamin N therapy group - metropolitan park environment (Experimental): Group with periodic outings to a neighborhood or metropolitan natural park (once a week) for approximately 2 hours for a minimum period of six months.
  Interventions: Other: Immersion therapy in nature - Vitamin N
- Group 2B: Vitamin N therapy group - forest forest environment (Experimental): Group with periodic outings to a forest environment (once a week) for a time of approximately 2 hours for a minimum period of six months
  Interventions: Other: Immersion therapy in nature - Vitamin N

INTERVENTIONS:
Other: Immersion therapy in nature - Vitamin N — Usual therapy group The first saliva sample will be taken upon awakening to determine cortisol concentration. At their workplace, they will be asked to remain seated and silent for 3 minutes, the following will be taken: blood pressure, heart rate, psychological instruments (stress-anxiety), blood sample.
  Group 2A and Group 2B In the natural environment, a saliva sample will be taken upon awakening to determine cortisol concentration. After arrival at the site, they will be asked to remain seated and silent for 3 minutes, the following will be taken: blood pressure, heart rate, psychological instruments (stress-anxiety), blood sample.
  The first phase is a session of observation of the site for 15 minutes. A slow, unhurried walk will be performed for 1 hour and 45 minutes. The order of activities (sitting and walking) will be established to ensure reliability of physiological measurements.
  Other Names: Shinrin-yoku
  Arms: Group 2A: Vitamin N therapy group - metropolitan park environment; Group 2B: Vitamin N therapy group - forest forest environment

SUMMARY:
Recent studies on health personnel in Colombia have evidenced the considerable increase in the levels of stress and anxiety, among other psychological disorders, as a product of the COVID-19 pandemic that is being experienced since 2019 and that implies a greater demand for attention from the affected citizens, with the consequent work overload and tension due to the risk of contagion.

Thus, the present work will allow the generation of new knowledge in relation to the benefits of Vitamin N therapy in Colombia; which can contribute quickly and effectively to the reduction of stress levels, anxiety, insomnia, and depression in individuals, when compared with conventional interventions and result in possible benefits such as the reduction of health problems such as obesity, diabetes, high blood pressure, and diseases associated with the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Persons over 18 years of age
* Health care workers
* Prioritized by the psychosocial risk program
* Complete vaccination schedule for COVID-19

Exclusion Criteria:

* Undergraduate students in the area of health sciences
* Pregnant women
* Allergies or sensitivity to the intervention
* Workers who consume immunosuppressants or corticosteroids
* Workers diagnosed with any type of disease or who have undergone chemotherapy or radiotherapy treatment during the last year
* Persons who have had exposure to X-rays in the last 6 months

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of Cortisol in saliva | 1 time per month for 6 months
  Saliva samples from each subject will be obtained with the Salivette device during each day of the intervention.
Outcome Measures in Arterial pressure levels | 4 time per month for 6 months
  Blood pressure in mm Hg before and after surgery
Outcome Measures in Heart rate levels | 4 time per month for 6 months
  Determination by digital sphygmomanometers
Change Psychological stress measurement scale levels | Three times for 6 months
  Determination of a score of the level of occupational stress through different

SECONDARY OUTCOMES:
Natural Killer | 1 time per month for 6 months
  Proportion of natural killer cells by flow cytometry.
Beck Anxiety Inventory levels | Three times for 6 months
  Determination of a score of the level of anxiety through different items taken into account in this instrument.
NR3C1 and FKBP5 gene methylation. | Two times for 6 months
  Percentage of methylation of NR3C1 and FKBP5 genes.
Pittsburgh Sleep Quality levels | Three times for 6 months
  Determination of a sleep quality score through different items taken into account in this instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Salud, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No